CLINICAL TRIAL: NCT06124651
Title: Clinical Comparison of Cruciate Retaining and Posterior Stabilized Total Knee Arthroplasty in Same Patients
Brief Title: Comparison of Cruciate Retaining and Posterior Stabilized Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: tka_cr_ps
Record Dates: First submitted 2023-08-23; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis, Knee; Arthropathy of Knee Joint
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CR knee (Active Comparator): This type of total knee arthroplasty retains the posterior cruciate ligament.
  Interventions: Procedure: Total knee replacement with cruciate retaining femoral component
- PS knee (Active Comparator): This type of total knee sacrifices the posterior cruciate ligament and cam and post mechanism replaces its function.
  Interventions: Procedure: Total knee replacement with cruciate substituting femoral component

INTERVENTIONS:
Procedure: Total knee replacement with cruciate retaining femoral component — To perform the total knee replacement, the knee joint is anatomically dissected, and thin portions of bone and cartilage is resected to accommodate a metallic implants. Implants are fixed to patients' bone with bone cements. Many designs for femoral component designs are available. In the present study, two types of implants, one CR(cruciate retaining), where the posterior cruciate ligaments are retained, and one PS(Posterior cruciate substituting), where the posterior cruciate ligaments are resected, will be compared. To make the comparison more reliable, the same kind of implants will be used, so that the major portions of femoral component design remains the same and the tibial component remains the same. Only the cruciate ligament parts are different. For this arm of intervention, CR knee will be used, so posterior cruciate will remain intact after the surgery and still function to aid in the knee stability.
  Arms: CR knee
Procedure: Total knee replacement with cruciate substituting femoral component — To perform the total knee replacement, the knee joint is anatomically dissected, and thin portions of bone and cartilage is resected to accommodate metallic implants that has similar contours of a native knee. Implants are fixed to patients' bone with bone cements. This procedure will use the femoral component that sacrifice the posterior cruciate ligament and having a box area with a post, so that "cam-post" mechanism of implants can mimic the function of the posterior cruciate ligament. To make the comparison more reliable, the same kind of implants will be used, so that the major portions of femoral component remains the same. The tibial component will remain the same design. Therefore, only the cruciate ligament parts will be different.
  Arms: PS knee

SUMMARY:
Several authors and large registries have suggested the potential for an increased risk of all-cause revision with the use of posterior cruciate-substitution (PS) total knee arthroplasty (TKA). The purpose of the current study was to compare posterior cruciate retaining (CR) and PS implants with respect to the functional and radiographic results, prevalence of osteolysis, revision rates and survivorship.

DETAILED DESCRIPTION:
The supremacy debate between posterior cruciate-retaining (CR) and posterior stabilized (PS) total knee arthroplasty (TKA) has now entered into the 4th decade. Multiple research studies have investigated CR and PS TKAs on the basis of kinematic, clinical, radiographic, and survivorship analysis. Despite arguments in favor of CR or PS TKA designs, several short or mid-term studies have shown no difference in functional outcomes between these two designs. Considering the fact that CR and PS TKA fare equally at short-term and mid-term, the decision to select either design should depend on their long-term survivorship. There have been few long-term survivorship analysis that have directly compared CR and PS TKAs with aseptic revision for any reason as the end point.

These long-term studies of CR and PS TKA have been done independently. A comparison of the results in the same patients eliminates the variability that is introduced by differences in gender, age, weight, comorbidity, bone quality, and activity level and allows for a meaningful comparison of the impact of fixation on the outcome of TKA. However, variability in terms of the preoperative severity of arthritis cannot be eliminated because of the design on both sides is rarely identical.

The purpose of this study was to identify differences in implant survivorship between CR and PS TKAs in patients with osteoarthritis who were younger than 65 years of age and CR implant in one knee and PS implant in the other.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee joint requiring total knee arthroplasty with bilateral disease

Exclusion Criteria:

* Inflammatory disease
* patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery
* Patient not medically cleared for bilateral surgery

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2006-06-30 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Improvement in Knee Society Knee Score | Initial(one day before surgery), at 3 months after the surgery, 1 year after the surgery, and then average 1 year after until the study completion
  change in knee score will be compared with initial score, until mean follow up of 25 years. The score ranges from 0 to 100, and the 100 is the highest.

SECONDARY OUTCOMES:
Improvement in the Range of motion | Initial(one day before surgery), and at 3 months after the surgery, 1 year after the surgery, and then average 1year after surgery until the study completion.
  change in the range of motion of knee joint will be compared with the initial value, until mean follow up of 25 years.The range of motion for knee typically are around 0 degrees to 130 degrees, and more range is considered as a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Young Hoo Kim, MD, Principal Investigator — Professor